CLINICAL TRIAL: NCT01266525
Title: A Multinational, Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled Study of the Effect on Cognitive Performance, Safety, and Tolerability of SAR110894D at the Doses of 0.5 mg, 2 mg, and 5 mg/Day for 24 Weeks in Patients With Mild to Moderate Alzheimer's Disease on Stable Donepezil Therapy
Brief Title: Effect of Different Doses of SAR110894 on Cognition in Patients With Mild to Moderate Alzheimer's Disease on Donepezil
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRI10734; 2010-022596-64 (EudraCT Number); U1111-1115-7535 (Other: UTN)
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Dementia Alzheimer's Type
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SAR110894 - 0.5 mg (Experimental): SAR110894, 0.5 mg once daily along with Donepezil.
  Interventions: Drug: SAR110894; Drug: Donepezil
- SAR110894 - 2 mg (Experimental): SAR110894, 2 mg once daily along with Donepezil.
  Interventions: Drug: SAR110894; Drug: Donepezil
- SAR110894 - 5 mg (Experimental): SAR110894, 5 mg once daily along with Donepezil.
  Interventions: Drug: SAR110894; Drug: Donepezil
- Placebo (Placebo Comparator): Placebo (for SAR110894) once daily along with Donepezil.
  Interventions: Drug: placebo (for SAR110894); Drug: Donepezil

INTERVENTIONS:
Drug: SAR110894 — Pharmaceutical form: Capsule
  Route of administration: Oral
  Arms: SAR110894 - 0.5 mg; SAR110894 - 2 mg; SAR110894 - 5 mg
Drug: placebo (for SAR110894) — Pharmaceutical form: Capsule
  Route of administration: Oral
  Arms: Placebo
Drug: Donepezil — 5 mg or 10 mg once daily continued as taken before inclusion

SUMMARY:
Primary Objective:

- To demonstrate the efficacy of at least one dose of SAR110894 (H3 receptor antagonist) in comparison to placebo on cognitive performance in patients with mild to moderate Alzheimer's disease (AD) while on stable donepezil therapy

Secondary Objectives:

* To explore the effect of SAR110894 on functional impairment, global clinical status and behavioral disturbances;
* To assess the safety/tolerability of SAR110894;
* To assess pharmacokinetic (PK) of SAR110894 and concentrations of donepezil;
* To explore caregiver time consumption and distress changes.

DETAILED DESCRIPTION:
The total study duration for each patient is approximatively 36 - 38 weeks broken down as follows:

* Screening period: up to 4 weeks,
* Treatment period: 24 weeks,
* Follow-up period: 10 weeks.

ELIGIBILITY:
Inclusion criteria:

* Patients with diagnosis of Alzheimer's Disease (AD) (Cannot be dementia from strokes or other causes).
* Patient is on stable and well-tolerated donepezil treatment at a dose of either 5 or 10 mg daily for at least 3 months prior to screening visit.

Exclusion criteria:

* Age <55 years old.
* Psychotic features, agitation, or behavioral problems within the last 3 months.
* Patients unable to comply with ophthalmologic monitoring.
* Lack of consistent and reliable caregiver.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2011-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Week 24 in the standard 11-item total score from the 13-item Alzheimer's Disease Assessment Scale - Cognitive subscale (ADAS-Cog). | Week 4, 12, and 24

SECONDARY OUTCOMES:
Change from baseline in the Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) global score | Week 4, 12, and 24
Change from baseline in each of the two remaining items of the ADAS-Cog (namely "delayed word recall" and "concentration/distractibility") | Week 4, 12, and 24
Change from baseline in each of the five factors from the Cognitive Drug Research System (CDR-S) computerized assessment | Week 4, 12, and 24
Change from baseline in the Mini Mental State Examination (MMSE) total score | Week 4, 12, and 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (82):
- United States (27):
  - Investigational Site Number 840041, Gilbert, Arizona
  - Investigational Site Number 840032, Phoenix, Arizona
  - Investigational Site Number 840024, Costa Mesa, California
  - Investigational Site Number 840013, Fresno, California
  - Investigational Site Number 840030, La Jolla, California
  - Investigational Site Number 840001, Redlands, California
  - Investigational Site Number 840002, Santa Ana, California
  - Investigational Site Number 840026, Sherman Oaks, California
  - Investigational Site Number 840034, Darien, Connecticut
  - Investigational Site Number 840003, Delray Beach, Florida
  - Investigational Site Number 840015, Hialeah, Florida
  - Investigational Site Number 840004, Jacksonville, Florida
  - Investigational Site Number 840006, Miami, Florida
  - Investigational Site Number 840012, Orlando, Florida
  - Investigational Site Number 840011, Tampa, Florida
  - Investigational Site Number 840005, West Palm Beach, Florida
  - Investigational Site Number 840008, Baton Rouge, Louisiana
  - Investigational Site Number 840025, Quincy, Massachusetts
  - Investigational Site Number 840009, Hattiesburg, Mississippi
  - Investigational Site Number 840040, Eatontown, New Jersey
  - Investigational Site Number 840018, Cedarhurst, New York
  - Investigational Site Number 840039, Charlotte, North Carolina
  - Investigational Site Number 840037, Tulsa, Oklahoma
  - Investigational Site Number 840014, Franklin, Tennessee
  - Investigational Site Number 840038, Austin, Texas
  - Investigational Site Number 840021, Bennington, Vermont
  - Investigational Site Number 840031, Williamsburg, Virginia
- Australia (9):
  - Investigational Site Number 036002, Adelaide
  - Investigational Site Number 036007, Chermside
  - Investigational Site Number 036008, Heidelberg West
  - Investigational Site Number 036006, Herston
  - Investigational Site Number 036001, Nedlands
  - Investigational Site Number 036004, Randwick
  - Investigational Site Number 036009, Toowoomba
  - Investigational Site Number 036005, Waratah
  - Investigational Site Number 036003, Woodville
- Canada (12):
  - Investigational Site Number 124010, Calgary
  - Investigational Site Number 124015, Gatineau
  - Investigational Site Number 124009, Greenfield Park
  - Investigational Site Number 124014, Halifax
  - Investigational Site Number 124001, London
  - Investigational Site Number 124011, Montreal
  - Investigational Site Number 124008, Ottawa
  - Investigational Site Number 124013, Regina
  - Investigational Site Number 124003, Sherbrooke
  - Investigational Site Number 124006, St. John's
  - Investigational Site Number 124002, Toronto
  - Investigational Site Number 124004, Toronto
- France (9):
  - Investigational Site Number 250004, Bordeaux
  - Investigational Site Number 250001, Lille
  - Investigational Site Number 250009, Limoges
  - Investigational Site Number 250007, Marseille
  - Investigational Site Number 250003, Nantes
  - Investigational Site Number 250005, Nice
  - Investigational Site Number 250006, Paris
  - Investigational Site Number 250008, Strasbourg
  - Investigational Site Number 250002, Toulouse
- Germany (6):
  - Investigational Site Number 276011, Berlin
  - Investigational Site Number 276012, Dresden
  - Investigational Site Number 276007, München
  - Investigational Site Number 276008, München
  - Investigational Site Number 276001, Schwerin
  - Investigational Site Number 276009, Würzburg
- Italy (6):
  - Investigational Site Number 380006, Ancona
  - Investigational Site Number 380004, Castellanza
  - Investigational Site Number 380005, Cefalù
  - Investigational Site Number 380002, Milan
  - Investigational Site Number 380001, Milan
  - Investigational Site Number 380003, Milan
- Poland (6):
  - Investigational Site Number 616004, Bydgoszcz
  - Investigational Site Number 616003, Gdansk
  - Investigational Site Number 616001, Gdynia
  - Investigational Site Number 616002, Poznan
  - Investigational Site Number 616006, Szczecin
  - Investigational Site Number 616005, Warsaw
- Portugal (2):
  - Investigational Site Number 620002, Amadora
  - Investigational Site Number 620001, Lisbon
- Spain (5):
  - Investigational Site Number 724002, Algorta
  - Investigational Site Number 724001, Barcelona
  - Investigational Site Number 724008, Madrid
  - Investigational Site Number 724007, Seville
  - Investigational Site Number 724003, Terrassa

REFERENCES:
- [Derived] McCleery J, Sharpley AL. Pharmacotherapies for sleep disturbances in dementia. Cochrane Database Syst Rev. 2020 Nov 15;11(11):CD009178. doi: 10.1002/14651858.CD009178.pub4. PMID 33189083
- [Derived] Leger D, Elbaz M, Dubois A, Rio S, Mezghiche H, Carita P, Stemmelin J, Strauss M. Alzheimer's Disease Severity is Not Significantly Associated with Short Sleep: Survey by Actigraphy on 208 Mild and Moderate Alzheimer's Disease Patients. J Alzheimers Dis. 2017;55(1):321-331. doi: 10.3233/JAD-160754. PMID 27662321